CLINICAL TRIAL: NCT06958744
Title: Effects of Functional Inspiratory Muscle Training on Diaphragm Function and Core Stabilization in Patients With Chronic Non-Specific Low Back Pain
Brief Title: Effects of Functional Inspiratory Muscle Training in Patients With Chronic Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, HATİCE HÜMEYRA AKIL, lecturer, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UUFTR01
Record Dates: First submitted 2025-04-19; First posted 2025-05-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Population Groups; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Inspiratory Muscle Training (FIMT) group (Experimental): Training will be given with the Powerbreath inspiratory muscle training device. Unlike traditional inspiratory muscle training, the exercises given in FIMT aim to integrate the functional capacity of respiratory muscles into daily life activities and include dynamic exercises in different positions with variable resistances. In this respect, it is defined as functional. Preparatory training will be given 4 weeks before starting FIMT: participants will be taught basic respiratory muscle training, respiratory control and exercises, and will be taught to perform the exercises while maintaining the spine in a neutral position. Patients will then be taken to FIMT for 3 days/6 weeks with a physiotherapist. On the other 3 days of the week, only inspiratory muscle training will be performed. The intensity of inspiratory muscle training will be increased from mild to moderate (Mild: Effort level between 20-40% of MIP or between Borg 2-3, Moderate: 50-60% of MIP or Borg 4-6).
  Interventions: Other: Functional Inspiratory Muscle Training (FIMT) group
- Control group (Active Comparator): Thoracic expansion exercise will be performed for 10 weeks. The participant will be asked to practice 4 times a day as a home program.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Functional Inspiratory Muscle Training (FIMT) group — Training will be given with the Powerbreath inspiratory muscle training device. Unlike traditional inspiratory muscle training, the exercises given in FIMT aim to integrate the functional capacity of respiratory muscles into daily life activities and include dynamic exercises in different positions with variable resistances. In this respect, it is defined as functional. Preparatory training will be given 4 weeks before starting FIMT: participants will be taught basic respiratory muscle training, respiratory control and exercises, and will be taught to perform the exercises while maintaining the spine in a neutral position. Patients will then be taken to FIMT for 3 days/6 weeks with a physiotherapist. On the other 3 days of the week, only inspiratory muscle training will be performed. The intensity of inspiratory muscle training will be increased from mild to moderate (Mild: Effort level between 20-40% of MIP or between Borg 2-3, Moderate: 50-60% of MIP or Borg 4-6).
  Arms: Functional Inspiratory Muscle Training (FIMT) group
Other: Control group — Thoracic expansion exercise will be performed for 10 weeks. The participant will be asked to practice 4 times a day as a home program.
  Arms: Control group

SUMMARY:
The aim of the study was to investigate the effects of functional respiratory muscle training on diaphragm function, core stabilization, respiratory muscle strength, pain, functional status and quality of life in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
Patients with chronic non-specific low back pain (CNSBP) have imbalances in postural control and kinetic chain. Postural control and respiratory function are mechanically and neuromuscularly interdependent. The diaphragm is the primary muscle in active inspiration with a vital role in contributing to spinal stability by modulating intra-abdominal pressure. The attachment of the diaphragm to the lumbar spine creates a synergistic working pattern with the transversus abdominis muscle. Altered activation patterns of the diaphragm and transversus abdominis have been observed in patients with chronic low back pain. Therefore, diaphragm function and respiratory pattern play a critical role in achieving and maintaining core stabilization. Studies have supported that different respiratory exercise programs are effective in reducing pain intensity, improving respiratory function and quality of life in CNSBP. These studies suggest a possible link between respiratory function, respiratory pattern, core stability and low back pain.

Inspiratory muscle training (IMT) is a technique used to increase the strength or endurance of the diaphragm and auxiliary respiratory muscles with a pressure threshold device. IMT consists of exercises involving breathing against resistance to improve respiratory muscle strength and aerobic capacity in healthy and sick populations. Respiratory muscles are also trunk muscles and their performance cannot be sufficiently optimized when respiratory muscle training is performed in isolation. Furthermore, if the load on the diaphragm, which has inspiratory, postural control and trunk stabilization tasks, increases, the muscle prefers breathing over these tasks. Functional training of the respiratory muscles is therefore recommended for optimal performance of the respiratory muscles. Functional inspiratory muscle training (FIMT) is defined as inspiratory respiratory muscle training during exercises in specific body positions. FIMT stimulates both the respiratory system and the core stabilization muscles as it consists of trunk and lumbopelvic exercises with stabilization of the spinal region during inspiratory load. Compared to traditional inspiratory muscle training, FIMT has a greater effect because it improves two roles of respiratory muscles (ventilation and spinal stabilization).

This study will investigate the effects of functional inspiratory muscle training (FIMT) on diaphragm thickness and mobility, respiratory muscle strength, core stabilization, pain, quality of life and functional status in patients with CNSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain lasting at least 3 months
* Being between the ages of 18 and 55
* Scoring 4 or more on the Numeric Pain Scale for the severity of low back pain
* Having a non-specific origin (not caused by a specific pathology such as -Infection, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome)
* Individuals with inspiratory muscle strength ≥80 mmHg
* Individuals with a forced expiratory volume (FEV1) of 80% or more

Exclusion Criteria:

* Tumor history
* Spine surgery in the last 12 months
* Spinal pathology (spondylolysis or spondylolisthesis) or concomitant neurological disease or neurological findings in the leg
* Having a chronic systemic disease
* Pregnancy
* Having a disease that affects the lungs and causes breathing problems
* Participation in a physiotherapy program in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Diaphragm Thickness | 10 weeks
  Diaphragm thickness (millimeter-mm) will be measured in the supine position with ultrasonography.

SECONDARY OUTCOMES:
The Numeric Rating Scale | 10 weeks
  NRS is a pain screening tool, used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Chest wall expansion | 10 weeks
  Chest wall mobility measurements will be taken at the axillary, xiphoid process and subcostal areas to assess chest wall mobility.
Respiratory muscle strength | 10 weeks
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements will be used to assess respiratory muscle strength.
McGill Core Endurance Test | 10 weeks
  Trunk muscle endurance tests developed by McGill include Sorensen test, trunk flexion, trunk extension, right-left lateral bridge test.
The Oswestry Disability Index | 10 weeks
  The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. The questionnaire examines the level of disability in 10 everyday activities of daily living. Each item consist of 6 statements which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest then the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.
36-Item Short Form Survey (SF-36) | 10 weeks
  It is used for objective measurement of quality of life. It comprises 36 questions that cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
Diaphragm Mobility | 10 weeks
  Diaphragm Mobility (millimeter-mm) will be measured in the supine position with ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Eyüboğlu, Principal Investigator — Uskudar University
Locations (1):
- Faculity of Health Sciences, Uskudar University, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No